CLINICAL TRIAL: NCT00676026
Title: The Impact of GABA-Enhancing Agents on Cortical GABA Concentrations Across the Menstrual Cycle in Women
Brief Title: Impact of GABA-Enhancing Agents on Cortical GABA Concentrations Across the Menstrual Cycle in Women
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Pennsylvania (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: Single | Purpose: Other
Other Study IDs: 0505027759
Record Dates: First submitted 2008-04-07; First posted 2008-05-12 (Estimated); Results first posted 2017-06-01 (Actual); Last update posted 2017-06-01 (Actual); Status verified 2017-05

CONDITIONS: Healthy
Keywords: menses; women; healthy controls; Healthy females with regular menstrual cycles
MeSH Terms: interventions — Fluoxetine; Zolpidem; Progesterone

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (3):
- Zolpidem 1 (Experimental): Zolpidem will be administered twice to each participant; once in the follicular and luteal phases of the menstrual cycle.
  Interventions: Drug: Zolpidem
- Progesterone 2 (Experimental): Progesterone will be administered twice to each participant; once in both the follicular and luteal phases of the menstrual cycle.
  Interventions: Drug: Progesterone
- Fluoxetine 3 (Experimental): Fluoxetine will be administered twice to each participant; once in both the follicular and luteal phases of the menstrual cycle.
  Interventions: Drug: Fluoxetine

INTERVENTIONS:
Drug: Fluoxetine — Fluoxetine 20 mg by mouth in the follicular and luteal phase of the menstrual cycle per participant.
  Other Names: Prozac
  Arms: Fluoxetine 3
Drug: Zolpidem — Zolpidem 10 mg by mouth in the follicular and luteal phase of the menstrual cycle per participant.
  Other Names: Ambien
  Arms: Zolpidem 1
Drug: Progesterone — Progesterone 800 mg by mouth will be administered to each participant once in the follicular and luteal phases of the menstrual cycle.
  Other Names: Prometrium
  Arms: Progesterone 2

SUMMARY:
The goal of this series of challenge studies is to examine the impact of menstrual cycle phase on cortical GABA response to administration of agents with either direct (benzodiazepines) or indirect (progesterone, fluoxetine) GABA modulating properties. While the impact of these agents on cortical GABA levels in women with premenstrual dysphoric disorder (PMDD) is of interest, this study is designed primarily for those women without a psychiatric illness.

ELIGIBILITY:
Inclusion Criteria:

* Women ages 18-45 and able to give voluntary written informed consent;
* Regular menstrual periods of 24-35 days in length;
* Body mass index 18.5 to 30 kg/m2;
* No past or present DSM-IV psychiatric or substance dependence diagnosis by structured diagnostic interview (SCID-NP); no substance abuse history within the previous 2 years;
* Absence of mood symptoms across the menstrual cycle during one month of prospective daily ratings with the Daily Record of Severity of Problems (DRSP); the DRSP is based on the DSM-IV research criteria for premenstrual dysphoric disorder (PMDD) and has been used in numerous studies to confirm the presence or absence of significant premenstrual mood and behavioral difficulties;
* Must be willing and able to participate in at least three of the four challenge paradigms.

Exclusion Criteria:

* Medical, neurologic or cerebrovascular disorder (CVA, seizure disorder, etc.);
* Family history of first degree relative with an Axis I psychiatric or substance dependence disorder (excepting alcohol and nicotine) (per subject report);
* Current treatment with psychoactive medication;
* Diabetes controlled by means other than diet;
* Use of steroid contraceptives (any method involving hormones) within the previous 4 months;
* Habitual consumption of more than 7 alcoholic drinks per week or more than 2 drinks on any particular occasion; must be willing to abstain from alcohol consumption for 48 hours prior to each 1H-MRS scan;
* Implanted metallic devices.

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 8 (Actual)
Dates: Start 2005-05; Primary Completion 2009-02 (Actual); Study Completion 2009-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Cynthia N Epperson, MD, Principal Investigator — Yale University
Locations (1):
- Yale University School of Medicine; Yale Program for Women's Reproductive Behavioral Health, New Haven, Connecticut, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were recruited at an outpatient research facility located at Yale University in New Haven, CT.
Groups:
- All Participants: This study was conducted at Yale University almost two decades ago. Our group at the University of Pennsylvania only has very basic information about this study. This includes the number of participants, which was 8, and the fact that no adverse events occurred. Staff members at the University of Pennsylvania do not have access to any additional study data. The contact person who initially entered this study protocol information is no longer at the University of Pennsylvania and we are unable to contact for additional information.
Period: Overall Study
Arm/Group | All Participants
Started | 8
Completed | 8
Not Completed | 0

BASELINE CHARACTERISTICS:
Population: As far as we know, data was never analyzed for this study. We only know that 8 participants completed.
Groups:
- All Participants: This study was conducted at Yale University almost two decades ago. Our group at the University of Pennsylvania only has very basic information about this study. This includes the number of participants, which was 18, and the fact that no adverse events occurred. Staff members at the University of Pennsylvania do not have access to any additional study data. The contact person who initially entered this study protocol information is no longer at the University of Pennsylvania and we are unable to contact for additional information.
Arm/Group | All Participants
Number analyzed (Participants) | 0
Age, Continuous [unit: years] — Population: UPenn does not have access to the data collected for this study. We are only using the information entered in the protocol section for very basic details in the results section (i.e, number of participants completed). The original contact person for this protocol is not reachable.
Sex: Female, Male — Population: UPenn does not have access to the data collected for this study. We are only using the information entered in the protocol section for very basic details in the results section (i.e, number of participants completed). The original contact person for this protocol is not reachable.

OUTCOME MEASURES:

1. Primary Outcome: To Determine the Impact of GABA-A Receptor Agonists (Benzodiazepines, Allopregnanolone) and Other GABA-modulating Agents (Fluoxetine) on Cortical GABA Levels by Menstrual Cycle Phase as Measured Using 1H-MRS in Healthy Controls.
Description: This study was conducted at Yale University almost two decades ago. Our group at the University of Pennsylvania only has very basic information about this study. This includes the number of participants, which was 8, and the fact that no adverse events occurred. Staff members at the University of Pennsylvania do not have access to any additional study data. The contact person who initially entered this study protocol information is no longer at the University of Pennsylvania and we are unable to contact for additional information.
Time Frame: Each medication will be administered 2 times during a 1-month menstrual cycle.
Population: UPenn does not have access to the data collected for this study. We are only using the information entered in the protocol section for very basic details in the results section (i.e, number of participants completed). The original contact person for this protocol is not reachable.
Arm/Group | All Participants
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Time Frame: Entire study duration.
Arm/Group | All Participants
All-Cause Mortality (participants affected / at risk) | 0/8
Serious Adverse Events (participants affected / at risk) | 0/8
Other Adverse Events (participants affected / at risk) | 0/8

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No